CLINICAL TRIAL: NCT01064258
Title: Reliability of Automatic CPAP Devices. A Double Blind Dummy Controlled Phase 1 Study
Brief Title: Trial of Auto Continuous Positive Airway Pressure (CPAP)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Daniel Rodenstein MD, Cliniques universitaires Saint-Luc
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2007/30MARS/67
Record Dates: First submitted 2010-02-04; First posted 2010-02-08 (Estimated); Last update posted 2010-02-16 (Estimated); Status verified 2010-02

CONDITIONS: Obstructive Sleep Apnea
Keywords: treatment; CPAP; sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fixed CPAP (Active Comparator): subject will sleep with a fixed CPAP device at minimal pressure
  Interventions: Device: CPAP
- autoCPAP (Experimental): the subject will sleep connected to an autoCPAP device
  Interventions: Device: autoCPAP

INTERVENTIONS:
Device: CPAP — CPAP at 4 cm H2O
  Arms: fixed CPAP
Device: autoCPAP — autoCPAP working between 4 and 15 cm H2O
  Arms: autoCPAP

SUMMARY:
Background: In patients with obstructive sleep apnea, automatic continuous positive airway pressure machines (autoCPAP) are said to be capable of identifying various breathing abnormalities during sleep and to correct them by increasing progressively the positive pressure applied to the airway. Once breathing becomes normal, pressure slowly declines. AutoCPAP devices have never been tested in Phase I studies. The investigators hypothesised that normal breathing would not be recognised as such, and that pressure would increase even in a normal subject.

DETAILED DESCRIPTION:
Material and Methods: We will submit one normal (confirmed with two polysomnographies, PSG) subject to a double blind study. Pairs of PSG will be performed on successive days once a week, one night with a 4 cm water fixed pressure CPAP device, previously shown not to disturb the subject's sleep and breathing, the other night with one of five well known autoCPAP devices programmed to work between 4 and 15 cm H2O pressure. The same mask and headgear will be used throughout the study. The subject and the physicians reading the tracings will ignore which device is being used on which night.

ELIGIBILITY:
Inclusion Criteria:

* normal subject
* male and female
* age 18 to 65 years old

Exclusion Criteria:

* obstructive sleep apnea
* unable to sleep with a CPAP device

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2009-08; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
number of episodes of increases in applied positive pressure, duration of each episode, and maximal pressure attained | one night

SECONDARY OUTCOMES:
reasons for pressure increase and consequences of the increase on sleep continuity | one night

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Rodenstein, MD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium

REFERENCES:
- [Derived] Mwenge GB, Dury M, Delguste P, Rodenstein D. Response of automatic continuous positive airway pressure devices in a normal subject. Eur Respir J. 2011 Jun;37(6):1530-3. doi: 10.1183/09031936.00139510. No abstract available. PMID 21632834